CLINICAL TRIAL: NCT01368172
Title: Implementation and Evaluation of the New Physical Activity Guidelines for People With Spinal Cord Injury.
Brief Title: Physical Activity Guidelines for People With Spinal Cord Injury (SCI)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: Rick Hansen Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: HicksPAGs
Record Dates: First submitted 2011-06-06; First posted 2011-06-07 (Estimated); Last update posted 2014-04-08 (Estimated); Status verified 2014-04

CONDITIONS: Spinal Cord Injury
Keywords: spinal cord injury; physical activity; physical fitness
MeSH Terms: conditions — Spinal Cord Injuries; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Physical Activity Guidelines (Experimental): Participants randomized to this arm received training/guidance on following the physical activity guidelines for adults with spinal cord injury
  Interventions: Behavioral: Physical Activity Guidelines
- Control (No Intervention)

INTERVENTIONS:
Behavioral: Physical Activity Guidelines — Participants in the Physical Activity Guidelines Arm will be asked to participate in at least 20 minutes of moderate to heavy intensity aerobic activity 2 times per week as well as strength training exercises (moderate intensity) 2 times per week. The Control Arm will not be supervised to follow the physical activity guidelines
  Arms: Physical Activity Guidelines

SUMMARY:
The first evidence-based physical activity guidelines for people with spinal cord injury were released in March, 2011. This project will evaluate the implementation of the new physical activity guidelines in a community exercise setting in Hamilton, Ontario. The investigators hypothesize that persons who follow the guidelines will experience increased aerobic fitness and muscle strength. The investigators also hypothesize that participants will find the guidelines easy to follow and that their self-efficacy for participating in physical activity will be improved following the study period.

ELIGIBILITY:
Inclusion Criteria:

* adults with spinal cord injury who have been given clearance to exercise by their primary care physician (or healthcare team)

Exclusion Criteria:

* ventilatory support
* inability to voluntarily participate in upper body exercises
* inability to communicate in English
* ongoing infection
* unstable autonomic dysreflexia

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2011-07; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Physical Fitness | 4 months
  Peak VO2 tests will be done on a cycle ergometer to assess aerobic capacity/endurance, and peak strength will be measured on accessible weight-training equipment.

SECONDARY OUTCOMES:
Self-efficacy for achieving the physical activity guidelines | 4 months
  Assessed through questionnaire.
Adherence to physical activity guidelines | 4 months
  Assessed through enrolment records

CONTACTS AND LOCATIONS:
Overall Officials: Audrey Hicks, PhD, Principal Investigator — McMaster University
Locations (1):
- Centre for Health Promotion and Rehabilitation, McMaster University, Hamilton, Ontario, Canada